CLINICAL TRIAL: NCT02541630
Title: A Pilot Study of Big Mind for Veterans With PTSD
Brief Title: Big Mind for Veterans With PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Attempts to recruit eligible subjects revealed that it would not be possible to enroll adequate numbers. Thus- no subjects were enrolled.
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniela Solzbacher, MD, Resident Physician, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00069755
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: PTSD
Keywords: Mindfulness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Big Mind — mindfulness based intervention

SUMMARY:
A variety of mindfulness-based interventions, such as Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy have been shown to be beneficial for individuals experiencing mood and anxiety symptoms. The aim of this pilot study is to test the feasibility of using a similar intervention, known as Big Mind, for veterans with PTSD and other psychological symptoms.

Big Mind is a method of self-exploration that utilizes a voice dialog technique to help individuals see the world and themselves from a variety of perspectives. The investigators hypothesize that this process will increase mindfulness and decrease self-referential thinking, which is associated with negative affect.

To test the feasibility of using this method, veterans with PTSD will complete a four-week group Big Mind class with a total of four sessions. The investigators will use a single group design with pre and post-intervention measures to assess tolerability and acceptance of the intervention. Secondary outcome measures will evaluate symptom improvement and increased mindfulness.

If this project demonstrates that using this intervention for veterans with PTSD is feasible, then more rigorous clinical trials will be warranted.

DETAILED DESCRIPTION:
In recent years, interventions involving mindfulness have become increasingly popular as complementary mind-body therapeutic strategies for a variety of medical and psychiatric conditions.

Mindfulness has been described as a practice of focusing attention on moment-by-moment experience with an attitude of curiosity, openness and acceptance. In other words, practicing mindfulness is simply experiencing the present moment. During mindfulness, awareness is focused on external sensory inputs, internal sensations, such as proprioception and pain, as well as awareness of the internal workings of the mind.

Mindfulness originated in Buddhist spiritual practices. One of these is Zen, a traditional Buddhist approach that primarily involves the practice of developing mindfulness by way of seated meditation. Two secular mindfulness-based interventions that have been extensively studied are Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT). MBSR was developed by Dr. Jon Kabat-Zinn at the University of Massachusetts Medical Center as secular method to utilize Buddhist mindfulness in mainstream psychology and medicine. MBSR includes education about stress as well as training on coping strategies and assertiveness in addition to mindfulness. MBCT was developed by Zindel Segal, Mark Williams and John Teasdale. MBCT is based upon MBSR and combines the principles of cognitive therapy with those of mindfulness to prevent relapse of depression. MBCT, like MBSR, utilizes secular mindfulness techniques including seated meditation.

A very large literature now supports the effectiveness of MBSR for social anxiety disorder, generalized anxiety disorder, improved psychological functioning among individuals with medical disorders and pain. Evidence indicates that MBCT is beneficial for unipolar depression relapse prevention, generalized anxiety disorder, panic disorder, hypochondriasis and social phobia. The strongest evidence is for relapse prevention in unipolar illness. Finally, a recent review and meta-analysis specifically addressed the effectiveness of MBSR and MBCT (and similar interventions) for reducing symptoms of anxiety and depression. The authors concluded that mindfulness based therapy improves symptoms of anxiety and depression across a wide range of severity and even when these symptoms are associated with other disorders.

The mechanisms underlying the effectiveness of mindfulness interventions are incompletely understood. However, considerable evidence suggests these approaches decrease depression and anxiety, at least in part, by altering self-referential thinking. For example, increased self-focused thinking is associated with affective symptoms. Furthermore, there is strong evidence that a particular type of thinking about self contributes to dysphoria in general and unipolar depression. Specifically, analytical self-focused rumination (thinking analytically about self and symptoms) is maladaptive. This cognitive style is associated with overgeneral autobiographical memory, global negative self-judgments, greater negative future thinking and dysphoria. Furthermore, there is compelling evidence that ruminative self-focus is associated with both the severity and duration of depressive symptoms as well as relapse of illness. In contrast to analytic self-focus, mindfulness (or experiential self-focus) is adaptive. Therefore, interventions that increase mindfulness and/or decrease analytical self-referential ruminations may be effective for depressive and anxiety symptoms. In fact, studies indicate that mindfulness approaches do in fact exert benefit as a result of both increasing mindfulness and decreasing self-focused rumination. These interventions also promote additional cognitive changes that may help ameliorate symptoms. One of these is enhancing compassion specifically including patience and kindness directed toward the self. Self-compassion is a predictor of psychological health and increases in caring for one's self appear to contribute to the effectiveness of these interventions.

There is considerable evidence that MBSR and MBCT have broad spectrum antianxiety and antidepressant effects as well as generally enhance psychological functioning and pain tolerance. Nonetheless, these approaches are unlikely to be effective for all patients. Thus, there is a need to evaluate the potential effectiveness of other mindfulness interventions. Further, the effectiveness of MBSR and MBCT suggests that other mindfulness interventions may also be beneficial and that studies of alternative approaches are warranted. Finally, there is a compelling need to evaluate the use of mindfulness approaches as adjunctive interventions for veterans with posttraumatic stress disorder (PTSD). The purpose of this study is to pilot test the feasibility of using an alternative mindfulness approach, Big Mind for veterans with PTSD seeking complementary and alternative treatment at the George E. Wahlen VAMC.

Big Mind (BM), developed by Zen Master Dennis Genpo Merzel is a secular mindfulness and self-discovery intervention that integrates aspects of Zen practice with a voice-dialogue method. Voice-dialog is sometimes used as a therapeutic tool in western psychology. The BM process guides individuals to shift their perspective, particularly in regard to self-perception.

BM facilitates self-discovery by teaching participants to become aware of different aspects of their sense of self by giving voice to these separate components. In other words, BM facilitates becoming "mindful" or more aware of one's own cognitions and emotions. Aspects of self may be cognitive constructs, such as the "Controller," the "Skeptic," the "Self-Critic," the "Cheater" and "Doubt" or emotional states, such as "Fear," "Anger," "Joy" or "Compassion" or sensations, such as "Pain." During a BM session, participants develop self-awareness by speaking as specific component, or "voice" of self, such as "the voice of Fear." Temporarily assuming the identity of an aspect in principle allows in depth exploration of the cognitions and emotions associated with that particular construct. The investigators hypothesize that his process can be therapeutically useful because facets associated with negative traits (e.g. the Cheater) or unpleasant affect (Fear) may be partially repressed and unacknowledged by the self. Bringing disowned voices to light facilitates working with cognitions and emotions in a more constructive way. For example, when one experiences chronic symptoms of anxiety (fear), the tendency is to try to avoid or prevent the unpleasant emotion. However, "fear of the fear" actually increases the discomfort and may result in the adoption of maladaptive strategies, such as excessive substance use or avoidance. Further, "fear of fear" likely exacerbates anxiety by increasing the baseline level of fear and perpetuating a vicious cycle of fear leading to even greater fear. BM offers a unique approach by giving active voice to the fear. Thus, one is able to examine the fear closely and come to recognize that it is transient and not harmful. When one both allows and actively encourages the experience of fear, the "fear of fear" dissipates and more adaptive behavior strategies can be adopted.

The BM process teaches how to shift perspective, therefore providing a means to escape the cycle of repetitive self-criticism and unconscious behavioral patterns and emotional responses. This is accomplished by viewing one's thoughts and behaviors from a neutral standpoint rather than from an ego based or self-focused perspective. Becoming "mindful" of these patterns facilitates taking conscious control of cognitive and emotional responses rather than being controlled by them.

In addition to decreasing negative cognitions and emotions, the investigators also hypothesize that BM increases mindfulness and decreases the analytic self-referential thinking associated with depression and PTSD. One can become less attached one's self-concept as well as the overall importance of self. This change in perception decreases the need to think about self analytically and increases one's ability to experience life in the here and now (mindfully).

BM has been used extensively over the last decade as a method of spiritual self-discovery. However, it has not been used as a clinical intervention. Scientific studies have not been conducted with the exception of one published study which suggested effectiveness as a rapid spiritual intervention tool. This study also provided preliminary evidence that the BM process increases mindfulness and decreases depression and anxiety. Based on the evidence for other mindfulness interventions discussed above, the investigators hypothesize that an adjunctive BM group intervention will decrease PTSD, mood and anxiety symptoms as well as increase physical pain tolerance among veterans with PTSD.

The Big Mind intervention will be presented in a group format. There will be four group sessions (90 minutes per group) and sessions will occur once weekly. Groups will be held in a classroom or group room at the George E. Wahlen VAMC. The number of subjects per intervention will be 5 - 10. The intervention will be repeated until a maximum of 30 subjects have been enrolled. Subjects will be given homework assignments to complete between group sessions. Each session will include BM group practice and review of homework assignments.

Study participants will complete six instruments at three time points of assessment: 1) baseline assessment prior to session one; 2) mid-point assessment during the intervention (end of week 2) and 3) post-intervention (end of week 4).

Attendance and reports of adverse events will be collected throughout the intervention.

Subject feedback will be obtained post-intervention (end of week 4).

ELIGIBILITY:
Inclusion Criteria:

* male and female veterans with PTSD
* age 18 - 65
* ability to provide informed consent

Exclusion Criteria:

* diagnosis of any psychotic disorder
* psychotic symptoms secondary to a mood disorder or other condition
* diagnosis of cognitive impairment or dementia
* currently on facility suicide high-risk list
* pregnancy
* impaired decision-making capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Feasibility | 4 weeks
  The investigators will assess tolerability and acceptance of the intervention via subjective feedback from each participant at the end of week 4, and monitor drop out rates.

SECONDARY OUTCOMES:
Improvement of PTSD symptoms | 4 weeks
  Improvement of PTSD symptoms will be measured via PCL-5 questionnaire.
Increase in mindfulness | 4 weeks
  Increase in mindfulness will be measured via the Five Facet Mindfulness Questionnaire.
Improvement of depressive symptoms | 4 weeks
  Improvement of depressive symptoms will be measured via HAM-D rating scale for depression.
Improvement of anxiety | 4 weeks
  Improvement of anxiety will be measured via HAM-A rating scale for anxiety.
Improvement of sleep | 4 weeks
  Improvement of sleep will be measured via Sleep Scale from the Medical Outcomes Study.

CONTACTS AND LOCATIONS:
Locations (1):
- George E. Whalen VAMC, Salt Lake City, Utah, United States